CLINICAL TRIAL: NCT04406025
Title: Regional Anesthesia Practice in Greece and Depiction of the Effect of Educational Activities in This Respect
Brief Title: Regional Anesthesia Practice in Greece
Acronym: Regional-Annie
Status: Completed | Type: Observational
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Other Study IDs: 194/25-02-2020
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Questionnaire; Survey
Keywords: seminar; regional anesthesia practice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- participation in Regional Anesthesia Seminar: this group consists of anesthesiologists that have attended a Regional Anesthesia Seminar taking place once a year
  Interventions: Procedure: participation in Regional Anesthesia Seminar
- no participation in Regional Anesthesia Seminar: this group consists of anesthesiologists that have not attended a Regional Anesthesia Seminar taking place once a year
  Interventions: Procedure: no participation in Regional Anesthesia Seminar

INTERVENTIONS:
Procedure: participation in Regional Anesthesia Seminar — this group of anesthesiologists attended the Regional Anesthesia Seminar
  Groups: participation in Regional Anesthesia Seminar
Procedure: no participation in Regional Anesthesia Seminar — this group of anesthesiologists did not attend the Regional Anesthesia Seminar
  Groups: no participation in Regional Anesthesia Seminar

SUMMARY:
The purpose of this structured questionnaire is to provide useful insight on the practice of regional anesthesia in Greece and depict the result of educational efforts taking place in the country to expand the knowledge and practice of regional anesthesia in the country

ELIGIBILITY:
Inclusion Criteria:

* greek anesthesia practitioners

Exclusion Criteria:

* nurses
* operating department assistants
* surgeons

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the polulation will be anesthesiologists practicing in Greece
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
knowledge and practice of regional anesthesia techniques | one month
  this is a 36-item free-text questionnaire, aiming at assessing knowledge and practice of regional anesthesia amongst participants

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang J, Gao H. Regional anesthesia practice in China: a survey. J Clin Anesth. 2016 Nov;34:115-23. doi: 10.1016/j.jclinane.2016.03.071. Epub 2016 May 3. PMID 27687357
- [Background] Smith MP, Sprung J, Zura A, Mascha E, Tetzlaff JE. A survey of exposure to regional anesthesia techniques in American anesthesia residency training programs. Reg Anesth Pain Med. 1999 Jan-Feb;24(1):11-6. doi: 10.1016/s1098-7339(99)90159-1. PMID 9952089